CLINICAL TRIAL: NCT02518529
Title: An Open, Multi-centre Study to Determine the Tolerability, Safety and Antibody Response Resulting From G17DT at 250mcg at Weeks 0, 2 and 6 With a Booster of 125mcg or 250mcg Given to Patients With Stage I - III Gastric Cancer
Brief Title: Study to Assess Tolerability and Safety and Antibody Response to G17DT in Gastric Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Collaborators: PPD Development, LP (Industry); ChapelPharma Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC12
Record Dates: First submitted 2015-08-04; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — gastrin immunogen

ARMS (1):
- 250µg dose treatment (Experimental): Subjects were treated with a 250mcg/0.2ml G17DT injection at weeks 0, 2 and 6.
  Interventions: Biological: G17DT

INTERVENTIONS:
Biological: G17DT
  Other Names: Gastrimmune, Insegia, PAS

SUMMARY:
Open-label, multicenter study to assess 250µg/0.2ml G17DT injection at weeks 0, 2 and 6. At or after week 20 and up to and including week 44. Subjects who raised antibodies to G17DT were given an additional dose of 125µg/0.1ml or 250µg/0.2ml G17DT between weeks 20-44 (study duration 52 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients who had had curative resection for histologically confirmed Stage I, II, or III gastric carcinoma or carcinoma of the oesophagogastric junciton.
* Male or female patients over 18 years of age.
* Patients with a life expectancy of at least four months.
* Karnofsky index for performance status of >70%
* Patients must have given written informed consent.

Exclusion Criteria:

* Gastric or junctional surgery within three weeks of baseline (week 0) or gastric or junctional surgery anticipated in the study period.
* History of other malignant disease within the previous five years, except non-melanomatous skin cancer or in situ carcinoma of the uterine cervix.
* Previous use (within the six weeks prior to the screening visit of the study), concomitant use, or anticipated use (up to week 16), of chemotherapy or immunotherapy.
* Previous use (within the six weeks prior to the screening visit of the study), concomitant use, or anticipated use (up to week 16), of radiotherapy or any other anti-cancer therapy.
* Previous use (within the four weeks prior to the screening visit of the study), concomitant use, or anticipated use (up to week 16), of immunosuppressants, including systemic corticosteroids.
* Known immunodeficiency.
* Females who were pregnant, planning to become pregnant or lactating. Women, who in the opinion of the investigator were of child bearing potential, were to have a negative pregnancy test before study drug administration.
* Patients taking part in another study involving an investigational or licensed drug or device in the three months preceding enrolment or up to week 16 during this study.
* Previous G17DT treatment.
* Haematological indicators:

Haemoglobin <10.0g/dl Neutrophils < 2.0 x 109/l Platelets <100 x 109/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2001-02; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Measurable Gastrin-17 Antibody Titer | Up to Week 52

SECONDARY OUTCOMES:
Injection tolerability | Up to Week 52
  Subjects were monitored for injection site reactions and/or swelling at the injections site.
Overall Survival from date of randomization to death or end of study | Up to December 2002